CLINICAL TRIAL: NCT05424588
Title: Effects of a 4400 km Ultra-cycling Non-competitive Race and Related Training on Body Composition and Circulating Progenitors Differentiation
Brief Title: Physical and Cellular Effects of Ultra-cycling
Acronym: ULTRABCD
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Dr. Michele Braggio (Unknown); Dr.ssa Maria Teresa Valenti (Unknown); Dr.ssa Arianna Minoia (Unknown); Dr. Gianluigi Dorelli (Unknown); Dr. Mattia Cominacini (Unknown); Prof. Francesco Bertoldo (Unknown); Dr.ssa Jessica Bertacco (Unknown); Dr.ssa Tonia De Simone (Unknown); Prof.ssa Maria Grazia Romanelli (Unknown); Prof.ssa Monica Mottes (Unknown); Dr.ssa Lekhana Bhandary (Unknown)
Responsible Party: Principal Investigator, Luca Giuseppe Dalle Carbonare, Associate Professor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: ULTRANORD
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Endurance Training
Keywords: ultra-cycling; training; body composition; cell differentiation
MeSH Terms: interventions — Physical Examination; Exercise Test; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy male amateur Caucasian cyclists: Healthy male amateur Caucasian cyclists who attended the NC4000 4th edition underwent clinical evaluation, bioelectrical impedance analysis (BIA), cardiopulmonary exercise testing (CPET) and venipuncture for blood samples collection.
  Interventions: Diagnostic Test: clinical evaluation, bioelectrical impedance analysis (BIA), cardiopulmonary exercise testing (CPET) and venipuncture for blood samples collection

INTERVENTIONS:
Diagnostic Test: clinical evaluation, bioelectrical impedance analysis (BIA), cardiopulmonary exercise testing (CPET) and venipuncture for blood samples collection — Total body dual-energy X-ray absorptiometry (DEXA) was taken BN and AN to measure total (FM) and segmental fat (truncal FM), visceral adipose tissue (VAT) and lean mass (LM). Tetra-polar dual frequency BIA (InBody 120; Cerritos, USA) was used BPP, BN and AN to measure weight and to estimate FM, FFM, and MM. Impedance measurements were performed. CPET was carried out on a cycle ergometer with clip-on pedals. Blood samples were collected in the morning BPP, BN, AN. Biochemical parameters considered in this study were: ALT, AST, creatinine, 25-hydroxy vitamin D, total cholesterol, HDL, LDL, triglycerides concentrations. We isolated CPCs from heparinized blood, as previously reported (14). After the collection of peripheral blood mononuclear cells (PBMCs) by a gradient centrifugation. (15). Differentiating Human Skeletal muscle cells were cultured with or without pooled sera of participants at 5% final concentration. 146b and 34a miRNAs were extracted from PBMCs.

SUMMARY:
Background: NorthCape4000 (NC4000) is the most participated ultra-endurance cycling race.

Eight healthy male Caucasian amateur cyclists were evaluated: a) before starting the preparation period; b) in the week preceding NC4000 (after the training period); c) after NC4000 race, with the aim to identify the effects of ultra-cycling on body composition, aerobic capacity and biochemical parameters as well as on the differentiation of progenitor cells.

Methods: Bioelectrical impedance analysis (BIA) and dual energy x-ray absorptiometry (DEXA) assessed body composition; cardiopulmonary exercise test (CPET) evaluated aerobic capacity. Differentiation of circulating progenitor cells was evaluated by analyzing the modulation in the expression of relevant transcription factors. In addition, in vitro experiments were performed to investigate the effects of sera of NC4000 participants on adipogenesis and myogenesis. The effects of NC4000 sera on Sestrins and Sirtuin modulation and the promotion of brown adipogenesis in progenitor cells was investigated as well. Two-tailed Student's paired-test was used to perform statistical analyses.

Results: We observed fat mass decrease after training as well as after NC4000 performance; we also recorded that vitamin D and lipid profiles were affected by ultra-cycling. In addition, our findings demonstrated that post-NC4000 participant's pooled sera exerted a positive effect in stimulating myogenesis and in inducing brown adipogenesis in progenitor cells.

Conclusions: The training program and Ultra-cycling lead to beneficial effects on body composition and biochemical lipid parameters, as well as changes in differentiation of progenitor cells , with significant increases in brown adipogenesis and in MYOD levels.

ELIGIBILITY:
Inclusion Criteria:

* male amateur Caucasian cyclists who attended the NC4000 4th edition

Exclusion Criteria:

* any condition that might have altered performance or laboratory tests results

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eight healthy male amateur Caucasian cyclists (47,5±13,5 years) who attended the NC4000 4th edition.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Body composition | DEC 2020-SEP 2021
  Total body dual-energy X-ray absorptiometry (DEXA) was taken BN and AN to measure total (FM) and segmental fat (truncal FM), visceral adipose tissue (VAT) and lean mass (LM)
Cell differentiation | DEC 2020-SEP 2021
  possible association with commitment of circulating progenitors.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI, Verona, Italy

IPD SHARING:
Plan to Share IPD: No